CLINICAL TRIAL: NCT03968393
Title: Anticoagulation for Stroke Prevention In Patients With Recent Episodes of Atrial Fibrillation Occurring Transiently With Stress - The ASPIRE-AF Trial
Brief Title: Anticoagulation for Stroke Prevention In Patients With Recent Episodes of Atrial Fibrillation Occurring Transiently With Stress
Acronym: ASPIRE-AF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-ASPIREAF; 2023-509142-35-00 (EU CTIS Number); 2019-001336-62 (EudraCT Number)
Record Dates: First submitted 2019-03-22; First posted 2019-05-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Atrial Fibrillation
Keywords: Transient Atrial Fibrillation; Perioperative Atrial Fibrillation; Non-vitamin K Oral Anticoagulation; Noncardiac Surgery; PROBE Design; Medical Illness; Stress
MeSH Terms: conditions — Stroke; Atrial Fibrillation | interventions — apixaban; Dabigatran; edoxaban; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label clinical trial with blinded outcome assessment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-vitamin K oral anticoagulant (NOAC) (Experimental): Participants randomized to the intervention arm will be prescribed one of the following NOACs for the duration of follow-up, unless they are undergoing a procedure with an increased risk of bleeding, have an adverse event or low calculated creatinine clearance, or decide to discontinue their use.
  Interventions: Drug: Non-vitamin K oral anticoagulant (NOAC)
- No anticoagulation (No Intervention): Participants randomized to the control arm will not be prescribed an oral anticoagulant unless they develop a clear indication for one during follow-up (e.g., recurrent nonoperative AF). They can be newly prescribed or continue taking low dose aspirin or another single antiplatelet agent as per the protocol. This will be decided by the participant's physician.

INTERVENTIONS:
Drug: Non-vitamin K oral anticoagulant (NOAC) — Participants randomized to the intervention arm will be prescribed one of the following NOACs for the duration of follow-up: edoxaban 60 mg daily (dose reduction to 30 mg, if applicable), apixaban 5 mg twice daily (dose reduction to 2.5 mg, if applicable), dabigatran 110 mg twice daily, or rivaroxaban 20 mg daily (dose reduction to 15 mg, if applicable). The choice of NOAC will be left up to the participant's prescribing physician.
  Other Names: Apixaban; Dabigatran; Edoxaban; Rivaroxaban
  Arms: Non-vitamin K oral anticoagulant (NOAC)

SUMMARY:
Multinational, investigator-initiated study of oral anticoagulation versus no anticoagulation for the prevention of stroke and other adverse cardiovascular events in patients with transient atrial fibrillation occurring transiently with stress and additional stroke risk factors.

DETAILED DESCRIPTION:
ASPIRE-AF is a prospective, randomized, open-label trial of non-vitamin K oral anticoagulants (NOACs) versus no oral anticoagulation in patients with transient atrial fibrillation and additional stroke factors occurring transiently with stress. The primary objective is to assess the effects of NOACs versus no anticoagulation on the co-primary composite outcomes of 1. non-hemorrhagic stroke and systemic embolism, and 2. vascular mortality, and non-fatal non-hemorrhagic stroke, myocardial infarction, peripheral arterial thrombosis, amputation, and symptomatic venous thromboembolism over the duration of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. have ≥1 episode of clinically important AFOTS during any of the following conditions:

   1. noncardiac surgery in the past 35 days, with at least an overnight hospital admission aftersurgery;
   2. noncardiac day surgery resulting in a large enough physiological insult to be able to cause AFOTS, as judged by the local investigator; or
   3. acute medical illness requiring hospital admission in the past 35 days and resulting in a large enough physiological insult to be able to cause AFOTS, as judged by the local investigator;
2. sinus rhythm at the time of randomization;
3. any of the following high-risk criteria:

   1. age 55-64 years, and having either known cardiovascular disease, recent major vascular surgery, a CHA2DS2VASc score ≥3, or an elevated postoperative troponin level;
   2. age 65-74 years, and having either known cardiovascular disease, recent major vascular surgery, a CHA2DS2VASc score ≥2, or an elevated postoperative troponin level; OR
   3. age ≥75 years.;
4. provide written informed consent

Exclusion Criteria:

1. any cardiac diagnosis as the primary reason for hospital admission;
2. history of documented chronic AF prior to noncardiac surgery;
3. need for long-term systemic anticoagulation;
4. ongoing need for long-term dual antiplatelet treatment;
5. contraindication to oral anticoagulation;
6. severe renal insufficiency (CrCl <20 ml/min);
7. severe liver cirrhosis (i.e., Child-Pugh Class C)
8. acute stroke in the past 14 days;
9. underwent cardiac surgery in the past 35 days;
10. history of nontraumatic intracranial, intraocular, or spinal bleeding;
11. hemorrhagic disorder or bleeding diathesis;
12. expected to be non-compliant with follow-up and/or study medications;
13. known life expectancy less than 1 year due to concomitant disease;
14. women who are pregnant, breastfeeding, or of childbearing potential who are not taking effective contraception; OR
15. previously enrolled in the trial

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2270 (Estimated)
Dates: Start 2019-06-14 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Non-hemorrhagic stroke or systemic embolism | For the duration of follow-up, until final follow-up (occurs when the last global participant has been followed for 24 months)
Incidence of vascular mortality, and non-fatal non-hemorrhagic stroke, myocardial infarction, peripheral arterial thrombosis, amputation, and symptomatic venous thromboembolism | For the duration of follow-up, until final follow-up (occurs when the last global participant has been followed for 24 months)

SECONDARY OUTCOMES:
Incidence of vascular mortality | For the duration of follow-up, until final follow-up (occurs when the last global participant has been followed for 24 months)
Incidence of non-fatal, non-hemorrhagic stroke | For the duration of follow-up, until final follow-up (occurs when the last global participant has been followed for 24 months)
Incidence of Myocardial infarction | For the duration of follow-up, until final follow-up (occurs when the last global participant has been followed for 24 months)
Incidence of peripheral arterial thrombosis | For the duration of follow-up, until final follow-up (occurs when the last global participant has been followed for 24 months)
Incidence of amputation | For the duration of follow-up, until final follow-up (occurs when the last global participant has been followed for 24 months)
Incidence of symptomatic venous thromboembolism | For the duration of follow-up, until final follow-up (occurs when the last global participant has been followed for 24 months)
Incidence of all-cause stroke | For the duration of follow-up, until final follow-up (occurs when the last global participant has been followed for 24 months)
Incidence of all-cause mortality | For the duration of follow-up, until final follow-up (occurs when the last global participant has been followed for 24 months)

OTHER OUTCOMES:
Incidence of composite of life-threatening, major, and critical organ bleeding | For the duration of follow-up, until final follow-up (occurs when the last global participant has been followed for 24 months)
  Safety objective, measured as previously done in the MANAGE trial
Incidence of major bleeding | For the duration of follow-up, until final follow-up (occurs when the last global participant has been followed for 24 months)
  Safety objective, measured according to the ISTH criteria
Incidence of hemorrhagic stroke | For the duration of follow-up, until final follow-up (occurs when the last global participant has been followed for 24 months)
  Safety objective
Hospitalization for vascular causes | For the duration of follow-up, until final follow-up (occurs when the last global participant has been followed for 24 months)
  Tertiary Objective
Hospitalization for all causes | For the duration of follow-up, until final follow-up (occurs when the last global participant has been followed for 24 months)
  Tertiary Objective

CONTACTS AND LOCATIONS:
Overall Officials: David Conen, MD, MPH, Principal Investigator — Population Health Research Institute; PJ Devereaux, MD, PhD, Study Chair — Population Health Research Institute
Locations (105):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mcgovern Medical School at University of Texas, Houston, Texas
- Argentina (7):
  - Clinica Coronel Suarez, Coronel Suárez, Buenos Aires
  - Instituto de Investigaciones Clinicas Rosario, Rosario, Santa Fe Province
  - Instituto Cardiovascular de Rosario, Rosario, Santa Fe Province
  - Centro Integral de Arritmias de Tucuman (CIAT), San Miguel de Tucumán, Tucumán Province
  - Hospital Municipal Chivilcoy, Chivilcoy
  - Sanatorio Cisma, San Miguel de Tucumán
  - Hospital Privado de Rosario, Santa Fe
- Australia (14):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Bankstown Hospital, Bankstown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast Hospital and Health Service, Birtinya, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Northeast Health Wangaratta, Wangaratta, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Brazil (2):
  - Instituto do Coração do Hospital das Clínicas da FMUSP, Cerqueira César
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
- Canada (24):
  - Foothills Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Medicine Hat Regional Hospital, Medicine Hat, Alberta
  - East Kootenay Regional Hospital, Cranbrook, British Columbia
  - Fraser Health Authority, Surrey, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - Dr.-Georges-L.-Dumont University Hospital Centre, Moncton, New Brunswick
  - Halifax Infirmary, Halifax, Nova Scotia
  - Cape Breton University, Sydney, Nova Scotia
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - The Ottawa Hospital General Campus, Ottawa, Ontario
  - Niagara Health System - St. Catharine's Site, St. Catharines, Ontario
  - Cortelluci Vaughan Hospital, Vaughan, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - CHU de Quebec Universite Laval, Québec, Quebec
  - Hôpital Fleurimont du Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Regina General Hospital, Regina, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Hospital South West Jutland - University Hospital of Southern Denmark, Esbjerg
  - Odense University Hospital, Odense
- Southwest Finland Wellbeing County (VARHA), Turku, Finland
- Universitatsklinikum Leipzig, Leipzig, Germany
- India (10):
  - GNRC Medical, North Guwāhāti, Assam
  - Marengo CIMS Hospital, Ahmedabad, Gujarat
  - NU Hospitals, Bangalore, Karnataka
  - Govt. T.D. Medical College, Alappuzha, Kerala
  - Amala Institute of Medical Sciences, Thrissur, Kerala
  - Amala Institute, Thrissur, Kerala
  - St. John's Medical College Hospital, Bangalore
  - JIPMER, Puducherry
  - Ruby Hall Clinic, Pune
  - Trivandrum Medical, Thiruvananthapuram
- Italy (5):
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Milan
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico, Milan
  - La Maddalena, Palermo
  - Piacenza Ospedale, Piacenza
- Nepal (3):
  - Nobel Medical College Teaching Hospital, Biratnagar
  - B.P. Koirala Institute of Health Sciences, Koshi
  - B and B Hospital, Lalitpur
- Netherlands (12):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep, Alkmaar
  - ZiekenhuisGroepTwente (ZGT), Almelo
  - Ziekenhuis Amstelland, Amstelveen
  - Rijnstate Hospital, Arnhem
  - Amphia Ziekenhuis Breda, Breda
  - Deventer Ziekenhuis, Deventer
  - Hospital Gelderse Vallei, Ede
  - Martini Hospital, Groningen
  - Franciscus Gasthuis, Rotterdam
  - Ikazia Hospital, Rotterdam
  - ETZ Tilburg, Tilburg
- Pakistan (5):
  - Aga Khan University, Karachi, Sindh
  - Maroof International Hospital, Islamabad
  - Shifa International Hospital, Islamabad
  - Dow Medical University, Karachi
  - Rehman Medical Institute, Peshawar
- South Korea (3):
  - Korea Univesrity Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul National University Bundang Hospital, Seoul
- Spain (6):
  - Hospital de Mar, Barcelona, Barcelona
  - Vall d'Hebron Hospital, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Mutua de Terrassa, Barcelona
  - University Hospital Ramon y Cajal, Madrid
  - Hospital Universitario de Navarra, Pamplona
- Sweden (2):
  - Karolinska Institutet Danderyd Hospital, Danderyd
  - Uppsala University, Uppsala
- Switzerland (3):
  - University Hospital Basel, Basel, Basel
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
- United Kingdom (2):
  - Liverpool Heart and Chest Hospital, Liverpool
  - Southend Hospital, Westcliff-on-Sea

IPD SHARING:
Plan to Share IPD: Undecided